CLINICAL TRIAL: NCT03657303
Title: Functional Exercise Response on osteoArthritis Relaxation Imaging
Acronym: FERARI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Fiona J Gilbert, Head of Department - Radiology, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A094874
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis
Keywords: Joint Diseases; Musculoskeletal Diseases; Arthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Arthritis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers
  Interventions: Device: Magnetic resonance imaging (MRI)
- Osteoarthritis patients
  Interventions: Device: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: Magnetic resonance imaging (MRI) — Participants will undergo an initial (baseline) MR examination, followed by repeat MR examinations at approximately 1 month and 1 year following the baseline examination.

SUMMARY:
Osteoarthritis (OA) is the most prevalent cause of mobility impairment and disability in the elderly. Indications at early stages of OA include decreased organisation of the collagen matrix, loss of proteoglycans and increased hydration. Late-stage joint disease can be diagnosed with X-ray, CT, and conventional MRI, but there are no validated methods to image early changes in cartilage microstructure, which are direly needed in early phase clinical development. Newly developed therapies and evaluation techniques are required at earlier stages of disease to offset the growing numbers and costs of end-stage disease.

MRI can probe soft-tissue with physical measurements that are not available through other methods. Quantitative MRI signal relaxation properties are particularly promising for assessing early changes in the cartilage composition. These relaxation properties are sensitive to water content and cartilage macromolecular structure.

Mechanical joint-loading and exercise affects quantitative MRI through cartilage compression and nonuniform deformation. A study measuring MRI relaxation times and using static joint-loading weights has shown differences between OA and healthy subjects. Cartilage volume, which is expected to be related to these relaxation times, recovers within an hour after exercise in healthy runners, with the menisci lagging in their volume recovery rate. Previous exercise studies have not measured post-exercise cartilage recovery using compositional techniques, such as physiologically-sensitive T1ρ and T2, nor probed compositional responses with OA subjects.

The investigators will examine a single knee of an initial 18 participants with MR. Participants will be drawn from two groups: (1) 12 participants aged 40-60 years old with clinical and x-ray features of OA and (2) 6 control subjects (matched to cases for age, sex and body mass index in a 1:2 ratio) who do not have clinical features of OA.

Participants will undergo an initial (baseline) MR examination, followed by repeat MR examinations at approximately 1 month and 1 year following the baseline examination.

This will allow the investigators to explore the possibility of mechanical joint-loading and exercise to differentiate early stage OA from healthy subjects and assess both the reliability of the MR measurements and the expected progression in the MR measurements in OA subjects in the absence of any disease-modifying intervention.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* Meets ACR criteria for OA Kellgren-Lawrence grade 2-3 on knee radiograph
* Neutral alignment
* Single symptomatic joint
* Aged 40-60 years old
* Ambulatory and in good general health
* Knee able to fit inside in-vivo knee coil (approx. 18 cm diameter)

Group 2 Inclusion Criteria:

* No current symptoms of knee pain or stiffness or other clinical features of OA
* Aged 40-60 years old
* Written consent to participate in the study
* Ambulatory and in good general health
* Knee able to fit inside in-vivo knee coil (approx. 18 cm diameter)

Exclusion Criteria for both groups:

* History of ipsilateral lower limb fracture
* History of ipsilateral lower limb surgery (including arthroscopy)
* Metabolic bone disease
* Inflammatory arthritis
* Haematological malignancy
* Paget's disease
* Bone metastases
* Contraindication to MR imaging (e.g. pacemaker, severe claustrophobia)
* No pregnant patients will be included
* Unable to consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1 will consist of 12 patients aged 40-60 who have presented to the Orthopaedic clinic with a painful knee, and have mild/moderate OA on plain radiographs (Kellgren- Lawrence grade 2-3). Group 2 will consist of 5 healthy volunteer controls, matched (1:2 ratio) to cases for age, sex and body mass index who do not have knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Establish effect sizes for MR parameters in OA patients compared to healthy volunteers. | 1 year

SECONDARY OUTCOMES:
Establish effect sizes for MR parameters in subjects with OA at 1 year compared to baseline. | 1 year
Establish reliability of the MR protocol and analysis techniques. | 1 month - 1 year
  Test-Retest Reliability

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom